CLINICAL TRIAL: NCT01791400
Title: Study of Effects of Metoclopramide Versus Sumatriptan on Migraine Headache
Brief Title: Effect of Metoclopramide Versus Sumatriptan for Emergency Department Treatment of Migraine Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, Research Assistant, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-70
Record Dates: First submitted 2013-02-10; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Migraine Disorders
Keywords: Metoclopramide; Sumatriptan; migraine; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Metoclopramide; Sumatriptan; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sumatriptan (Other): Patients who underwent 6 mg sumatriptan subcutaneous one time
  Interventions: Drug: Sumatriptan, injection, 6 mg, one time
- Metoclopramide (Other): Patients who underwent 20 mg Metoclopramide intravenous one time
  Interventions: Drug: metoclopramide, injection,20mg, one time

INTERVENTIONS:
Drug: metoclopramide, injection,20mg, one time — metoclopramide, intravenous injection,20mg, one time
  Other Names: plasil
  Arms: Metoclopramide
Drug: Sumatriptan, injection, 6 mg, one time — Sumatriptan, subcutaneous injection, 6 mg, one time
  Arms: sumatriptan

SUMMARY:
The purpose of this study is to determine which drug makes lower migraine headache

DETAILED DESCRIPTION:
There are different options to manage benign headache in emergency department.The investigators compared Intravenous metoclopramide with Subcutaneous sumatriptan to relieve pain in emergency department.

ELIGIBILITY:
Inclusion Criteria:

* 20-60 years old and presented with acute headache similar to previous episodes,
* with or without phonophobia,
* photophobia,
* vomiting or nausea.

Exclusion Criteria:

* fever or neck stiffness,
* altered mental state,
* pregnancy,
* recent trauma or seizure (within 24 hours),
* focal neurological abnormality on physical examination,
* allergy to metoclopramide,
* hypertension,
* cardiovascular diseases.

Also if the patients had taken a triptan or ergot during the last 24 hours were excluded from the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
pain | at one hour after prescription
  determining pain in Metoclopramide versus sumatriptan groups

CONTACTS AND LOCATIONS:
Overall Officials: babak masoumi, A.Professor, Principal Investigator — Isfahan, Isfahan, Iran, Islamic Republic of
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran